CLINICAL TRIAL: NCT02413723
Title: McGrath Mac Videolaryngoscope Versus Macintosh Laryngoscope for Orotracheal Intubation in Critical Care Unit
Acronym: MACMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A00674-43
Record Dates: First submitted 2015-03-28; First posted 2015-04-10 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Intratracheal Intubation in Critical Care
Keywords: intubation; critical care; laryngoscope; videolaryngoscope; intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Videolaryngoscope McGrath Mac (Active Comparator): McGrath Mac videolaryngoscope will be used for laryngoscopy for patient's intubation
  Interventions: Device: Videolaryngoscope
- Standard laryngoscope (Placebo Comparator): Macintosh laryngoscope will be used for laryngoscopy for patient's intubation
  Interventions: Device: Standard laryngoscope

INTERVENTIONS:
Device: Videolaryngoscope — McGrath Mac videolaryngoscope will be use for first attempt of intratracheal intubation.
  Other Names: Mc Grath videolaryngoscope
  Arms: Videolaryngoscope McGrath Mac
Device: Standard laryngoscope — Macintosh laryngoscope will be use for first attempt of intratracheal intubation.
  Other Names: Macintosh laryngoscope
  Arms: Standard laryngoscope

SUMMARY:
The aim of this study is to demonstrate that the rate of successful orotracheal intubation at first laryngoscopy will be higher in patients intubated with McGrath Mac videolaryngoscope compared to patients intubated with classical Macintosh laryngoscope in patients requiring an orotracheal intubation in ICU.

ELIGIBILITY:
Inclusion Criteria:

• Requiring orotracheal intubation

Exclusion Criteria:

* Contraindication to orotracheal intubation
* Time too short to allow inclusion and randomisation of patient (particularly cardiac arrest)
* Minor (<18 )
* Pregnant, parturient , or breast-feeding woman
* Patient hospitalized without consent and/or deprived of liberty by court's decision
* Patient under guardianship or curators
* Lack of social insurance
* Lack of informed consent
* Concomitant inclusion in a trial whose primary endpoint focuses on intubation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proportion of successful orotracheal intubation at first laryngoscopy | intubation procedure, an expected average of 15 minutes
  Number of successful intubation at first laryngoscopy in one arm/number of included patients in the same arm.

SECONDARY OUTCOMES:
Proportion of successful orotracheal intubation all laryngoscopies pooled | intubation procedure, an expected average of 15 minutes
Time to successful orotracheal intubation | intubation procedure, an expected average of 15 minutes
  Defined by the time between the beginning of induction (injection of anesthetic drugs) and the time of confirmation of the intratracheal nature of the endotracheal tube (defined as apparition of first inflexion on the expired carbon dioxide curve)

OTHER OUTCOMES:
Cormack and Lehane grade | intubation procedure, an expected average of 15 minutes
Percentage of glottic opening (POGO) score | intubation procedure, an expected average of 15 minutes
Difficult Intubation | intubation procedure, an expected average of 15 minutes
Resort to alternative intubation technique | intubation procedure, an expected average of 15 minutes
Frequency of occurence of unexpected events | Discharge from Intensive Care unit, an expected average of 7 days
Mechanical ventilation duration | Time from extubation, an expected average of 6 days
Intensive Care Unit length of stay | Discharge from Intensive Care unit, an expected average of 7 days
Hospital length of stay | Discharge from hospital, an expected average of 14 days
Intensive Care Unit Mortality | Discharge from Intensive Care unit, an expected average of 7 days
Mortality at day 28 | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jean Baptiste Lascarrou, MD, Principal Investigator — CHD Vendee
Locations (7):
- France (7):
  - CHU Louis Mourier, Colombes
  - CHD Vendee, La Roche-sur-Yon
  - CHU Orleans, Orléans
  - CHU Saint Louis, Paris
  - CHU Paris Cochin, Paris
  - CHU Strasbourg Nouvel Hôpital Civil, Strasbourg
  - CHU Tours, Tours

REFERENCES:
- [Background] Lascarrou JB, Le Thuaut A, Reignier J. Intubation With Video Laryngoscopy vs Direct Laryngoscopy-Reply. JAMA. 2017 May 23;317(20):2131-2132. doi: 10.1001/jama.2017.4486. No abstract available. PMID 28535229
- [Background] Bailly A, Lascarrou JB, Le Thuaut A, Boisrame-Helms J, Kamel T, Mercier E, Ricard JD, Lemiale V, Champigneulle B, Reignier J; Clinical Research in Intensive Care and Sepsis Group. McGRATH MAC videolaryngoscope versus Macintosh laryngoscope for orotracheal intubation in intensive care patients: the randomised multicentre MACMAN trial study protocol. BMJ Open. 2015 Dec 23;5(12):e009855. doi: 10.1136/bmjopen-2015-009855. PMID 26700287
- [Result] Lascarrou JB, Boisrame-Helms J, Bailly A, Le Thuaut A, Kamel T, Mercier E, Ricard JD, Lemiale V, Colin G, Mira JP, Meziani F, Messika J, Dequin PF, Boulain T, Azoulay E, Champigneulle B, Reignier J; Clinical Research in Intensive Care and Sepsis (CRICS) Group. Video Laryngoscopy vs Direct Laryngoscopy on Successful First-Pass Orotracheal Intubation Among ICU Patients: A Randomized Clinical Trial. JAMA. 2017 Feb 7;317(5):483-493. doi: 10.1001/jama.2016.20603. PMID 28118659